CLINICAL TRIAL: NCT01781299
Title: Acellular Dermal Matrix in Tissue Expander Breast Reconstruction: A Prospective, Randomized, Clinical Trial Comparing SurgiMend PRS and AlloDerm RTU
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Ken Shestak, Principal Investigator, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRO11020226
Record Dates: First submitted 2013-01-24; First posted 2013-01-31 (Estimated); Results first posted 2017-05-12 (Actual); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Breast Cancer; Mastectomy
Keywords: Breast Cancer; Mastectomy; Immediate reconstruction
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: We are looking at 2 products called Acellular Dermal Matrix (ADM) implant to evaluate the outcomes of 2 specific ADM products: SurgiMend PRS and AlloDerm RTU.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AlloDerm RTU (Active Comparator): Participants within this arm will have the acellular dermal matrix AlloDerm RTU implanted at the time of tissue expander placement.
  Interventions: Device: AlloDerm RTU
- SurgiMend PRS (Active Comparator): Participants within this arm will have the acellular dermal matrix SurgiMend PRS implanted at the time of tissue expander placement.
  Interventions: Device: SurgiMend PRS

INTERVENTIONS:
Device: AlloDerm RTU
  Arms: AlloDerm RTU
Device: SurgiMend PRS
  Arms: SurgiMend PRS

SUMMARY:
The purpose of this study is to assess the relative performance and complication rates between the AlloDerm RTU and SurgiMend PRS products as well as the relative economics of these two treatment options.

DETAILED DESCRIPTION:
In recent years, acellular dermal matrix (ADM) products have increasingly been utilized in breast reconstruction in order to protect the implant from exposure under a thin mastectomy skin flap while also allowing better control of the inframammary fold and, therefore, a better cosmetic result. In current clinical practice, cost is a factor in considering procedures and adjunct products. AlloDerm RTU and SurgiMend PRS are dissimilar in cost, with AlloDerm RTU more costly by 30-50%, and it is unclear if they are similar in efficacy.

This study will be a prospective, randomized-to-test article (ADM), controlled, blinded-to-aesthetic/biopsy specimen evaluator trial. It will provide a way to assess the relative performance and complication rates between the AlloDerm RTU and SurgiMend PRS product as well as the relative economics of these two treatment options. Study subjects will only be randomized to one of two surgical mesh products. Patient information including age, BMI, smoking history, tumor size and location, preoperative bra cup size, mastectomy specimen weight, mastectomy method, plastic surgeon, mastectomy surgeon, quality of skin, tissue expander type and maximal volume, intra-operative fill volume, gel/saline implant type and size, chemotherapy, and radiation therapy will be summarized.

ELIGIBILITY:
Inclusion Criteria:

1. Subject's with ability to provide informed consent.
2. Subjects greater than 18 years old
3. Subjects to undergo an immediate tissue expander reconstruction following mastectomy; and
4. Subjects who are, in the opinion of the Investigator, able to understand the study, comply with the study design and are willing to return to the clinic for all the research required follow-up visits.

Exclusion Criteria:

1. Subjects less than 18 years of age
2. Subjects that based on surgeon's discretion cannot be effectively reconstructed with the use of ADM product
3. Pregnancy
4. Bovine allergy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Shestak, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Center for Innovation in Restorative Medicine, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Breuing KH, Warren SM. Immediate bilateral breast reconstruction with implants and inferolateral AlloDerm slings. Ann Plast Surg. 2005 Sep;55(3):232-9. doi: 10.1097/01.sap.0000168527.52472.3c. PMID 16106158
- [Background] Gamboa-Bobadilla GM. Implant breast reconstruction using acellular dermal matrix. Ann Plast Surg. 2006 Jan;56(1):22-5. doi: 10.1097/01.sap.0000185460.31188.c1. PMID 16374090
- [Background] Topol BM, Dalton EF, Ponn T, Campbell CJ. Immediate single-stage breast reconstruction using implants and human acellular dermal tissue matrix with adjustment of the lower pole of the breast to reduce unwanted lift. Ann Plast Surg. 2008 Nov;61(5):494-9. doi: 10.1097/SAP.0b013e31816d82d9. PMID 18948774
- [Background] Maxwell GP, Gabriel A. Possible future development of implants and breast augmentation. Clin Plast Surg. 2009 Jan;36(1):167-72, viii. doi: 10.1016/j.cps.2008.08.005. PMID 19055971
- [Background] Stump A, Holton LH 3rd, Connor J, Harper JR, Slezak S, Silverman RP. The use of acellular dermal matrix to prevent capsule formation around implants in a primate model. Plast Reconstr Surg. 2009 Jul;124(1):82-91. doi: 10.1097/PRS.0b013e3181ab112d. PMID 19568048
- [Background] Namnoum JD. Expander/implant reconstruction with AlloDerm: recent experience. Plast Reconstr Surg. 2009 Aug;124(2):387-394. doi: 10.1097/PRS.0b013e3181aee95b. PMID 19644253
- [Background] Grabov-Nardini G, Haik J, Regev E, Winkler E. AlloDerm Sling for Correction of Synmastia After Immediate, Tissue Expander, Breast Reconstruction in Thin Women. Eplasty. 2009 Nov 12;9:e54. PMID 20011582
- [Background] Sbitany H, Sandeen SN, Amalfi AN, Davenport MS, Langstein HN. Acellular dermis-assisted prosthetic breast reconstruction versus complete submuscular coverage: a head-to-head comparison of outcomes. Plast Reconstr Surg. 2009 Dec;124(6):1735-1740. doi: 10.1097/PRS.0b013e3181bf803d. PMID 19952627
- [Background] Nahabedian MY. AlloDerm performance in the setting of prosthetic breast surgery, infection, and irradiation. Plast Reconstr Surg. 2009 Dec;124(6):1743-1753. doi: 10.1097/PRS.0b013e3181bf8087. PMID 19952629
- [Background] Chun YS, Verma K, Rosen H, Lipsitz S, Morris D, Kenney P, Eriksson E. Implant-based breast reconstruction using acellular dermal matrix and the risk of postoperative complications. Plast Reconstr Surg. 2010 Feb;125(2):429-436. doi: 10.1097/PRS.0b013e3181c82d90. PMID 20124828
- [Background] Shatkin BT "A new option for implant-based breast reconstruction using SurgiMend PRS® (sterile, acellular bovine fetal dermis)" (in submission)
- [Background] Vinas, LA, Corbitt, JD, Anthony, L and Greenburg, AG "Fetal bovine acellular dermal matrix (SurgiMend PRS®) in one-stage immediate prosthetic breast reconstruction" (in submission)
- [Background] Lanier ST, Wang ED, Chen JJ, Arora BP, Katz SM, Gelfand MA, Khan SU, Dagum AB, Bui DT. The effect of acellular dermal matrix use on complication rates in tissue expander/implant breast reconstruction. Ann Plast Surg. 2010 May;64(5):674-8. doi: 10.1097/SAP.0b013e3181dba892. PMID 20395795
- [Background] Pusic AL, Klassen AF, Scott AM, Klok JA, Cordeiro PG, Cano SJ. Development of a new patient-reported outcome measure for breast surgery: the BREAST-Q. Plast Reconstr Surg. 2009 Aug;124(2):345-353. doi: 10.1097/PRS.0b013e3181aee807. PMID 19644246

RESULTS

PARTICIPANT FLOW:
Groups:
- AlloDerm RTU: Participants within this arm will have the acellular dermal matrix AlloDerm RTU implanted at the time of tissue expander placement.
  AlloDerm RTU
- SurgiMend PRS: Participants within this arm will have the acellular dermal matrix SurgiMend PRS implanted at the time of tissue expander placement.
  SurgiMend PRS
Period: Overall Study
Arm/Group | AlloDerm RTU | SurgiMend PRS
Started | 4 | 5
Completed | 4 | 4
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AlloDerm RTU | SurgiMend PRS | Total
Number analyzed (Participants) | 4 | 5 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 5 | 8
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (8.8) | 42 (3.9) | 48.7 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 5 | 8
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 5 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Complication Rates
Description: To determine the complication rate for tissue expander breast reconstruction patients using SurgiMend PRS and AlloDerm RTU ADM products. Time points include: After first procedure: 10-14 days, then 2, 4, 6, and 10 weeks after drain removal; After second procedure: 1-2 weeks, 6 weeks, 1 year, and 3 years.
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | AlloDerm RTU | SurgiMend PRS
Number analyzed (Participants) | 4 | 4
Participants | 4 | 3

2. Secondary Outcome: Aesthetic Evaluation
Description: Initial aesthetic evaluation will occur at approximately 6 weeks after permanent implant placement. Re-evaluation will occur at 1 and 3 years following permanent implant placement. This will involve physical examination, 2D photographs, and patient Breast-Q self-examination. Breast-Q examination is on a scale of 25-100 with 25 questions on a scale of 1-4 where 1 is very dissatisfied and 4 is very satisfied.
Time Frame: 3 years following permanent implant placement.
Population: discrepancy is caused by funding ending and no data was collected from SurgiMend arm.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | AlloDerm RTU | SurgiMend PRS
Number analyzed (Participants) | 2 | 0
units on a scale | 83.5 [83 to 84] |

ADVERSE EVENTS:
Arm/Group | AlloDerm RTU | SurgiMend PRS
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/5
Other Adverse Events (participants affected / at risk) | 0/4 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes